CLINICAL TRIAL: NCT03478293
Title: A Prospective Evaluation of the Second Generation iStent Inject in Open-Angle Glaucoma Subjects on Two Preoperative Topical Ocular Hypotensive Medications
Brief Title: iStent Inject in OAG Subjects on 2 Pre-op Topical Ocular Hypotensive Medications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-045
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Primary Open Angle Glaucoma (POAG)
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- iStent inject surgery (Experimental): Single-arm study. Intervention is micro-invasive glaucoma surgery (MIGS) to implant iStent inject
  Interventions: Device: iStent inject surgery

INTERVENTIONS:
Device: iStent inject surgery — Micro-invasive glaucoma surgery (MIGS) to implant iStent inject

SUMMARY:
The purpose of this study is to evaluate the intraocular pressure (IOP) lowering effect of iStent inject in eyes of subjects with primary open-angle glaucoma previously on two anti-glaucoma medications.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the intraocular pressure (IOP) lowering effect of iStent inject in eyes of subjects with primary open-angle glaucoma previously on two anti-glaucoma medications. Outcomes will be evaluated at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open angle glaucoma (POAG)
* Subject on two ocular hypotensive medications

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
IOP reduction at 12 and 24 months on same number or fewer medications | 12 months and 24 months
  IOP reduction at 12 and 24 months on same number or fewer medications

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, OD, Study Director — Glaukos Corporation
Locations (1):
- Department of Ophthalmology - UNIFESP/ Hospital São Paulo, São Paulo, Brazil